CLINICAL TRIAL: NCT06387628
Title: A Phase II Single Center Two Cohorts Trial of LM-108 in Combination With PD-1 Based Treatment for Patients With Recurrent or Metastatic Triple - Negative Breast Cancer
Brief Title: LM-108 in Combination With PD-1 Based Treatment for Patients With Recurrent or Metastatic Triple - Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LM108-IIT-202
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: TNBC - Triple-Negative Breast Cancer
Keywords: Immunotherapy; PD-1; CCR8; Triple-Negative Breast Cancer; TNBC
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — toripalimab; eribulin; Taxes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LM-108, toripalimab and eribulin (Experimental)
  Interventions: Drug: LM-108; Drug: Toripalimab; Drug: Eribulin
- LM-108, toripalimab and nab-paclitaxel (Experimental)
  Interventions: Drug: LM-108; Drug: Toripalimab; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: LM-108 — LM-108, 10mg/kg, d1, q6w
Drug: Toripalimab — Toripalimab, 240 mg, d1, q3w
Drug: Eribulin — Eribulin 1.4 mg/m2, d1, 8 , q3w
  Arms: LM-108, toripalimab and eribulin
Drug: Nab paclitaxel — Nab paclitaxel 125 mg/m2, d1, 8 , q3w
  Arms: LM-108, toripalimab and nab-paclitaxel

SUMMARY:
To evaluate the efficacy and safety of LM108 plus toripalimab plusnab-paclitaxel or eribulin as first-line or post-line treatment in patients with metastatic triple-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old (including boundary value), no gender limit;
2. ECOG score 0-1;
3. Expected survival ≥3 months;
4. Unresectable or metastatic or postoperative recurrent, histologically confirmed advanced triple-negative breast cancer. Triple-negative breast cancer is defined as: ER, PR and HER2 are negative. ER-negative and PR-negative are defined as tumors without positive staining, the proportion of cells in all tumor cells is <1%; HER2-negative is defined as: HER2 (0), HER2 (1+) or HER2 (2+) detected by immunohistochemistry but negative by fluorescence in situ hybridization (FISH); Cohort 2 requires histological confirmation of PD-L1 CPS ≥ 1;
5. Cohort 1 : at least one prior line at recurrence or metastasis setting with disease progression or intolerable toxicity. In this situation, patients are allowed to be enrolled: the time between the last intravenous dose of adjuvant chemotherapy and first recurrence or metastasis is ≤6 months. Cohort 2: no prior line at recurrence or metastasis setting is allowed, the time between the last intravenous dose of adjuvant chemotherapy and first recurrence or metastasis ≥12 months.;
6. Provide sufficient fresh tissue specimens for biomarker analysis before treatment;
7. According to RECISTv1.1 standard, there is at least 1 measurable lesion;
8. Appropriate bone marrow and organ function before first dose :

   * Bone Marrow: Platelets ( PLT ) ≥ 90 × 109 /L , absolute neutrophil count ( ANC ) ≥ 1.5 × 109 /L , hemoglobin ≥ 9 g/dL ;
   * Coagulation: INR ≤ 1.5 , APTT ≤ 1.5 × ULN ;
   * Liver function: Liver function is basically normal, total bilirubin ≤ 1.5 × ULN ( total bilirubin in patients with Gilbert syndrome ≤ 3 × ULN can be enrolled), AST and ALT ≤ 2.5 × ULN (if there is liver metastasis, AST , ALT ≤ 5 × ULN );
   * Renal function: serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min (according to Cockcroft-Gault formula);
   * Cardiac function: left ventricular ejection fraction ( LVEF ) ≥ 50% ; female QT interval ( QTcF ) ≤ 470 ms , male ≤ 450 ms .
9. Be able to well communicate with the investigator and understand and comply with the requirements of this study.

Exclusion Criteria:

1. Cohort 1 : Previous use of eribulin and CCR8- targeting drugs; Cohort 2: previous use of CCR8-targeting drugs and nab-paclitaxel, unless the interval between the last dose of nab-paclitaxel in the adjuvant chemotherapy and first recurrence or metastasis is ≥12 months;
2. Have received radiotherapy, chemotherapy, traditional Chinese medicine with anti-tumor indications, and local therapy (interventional therapy but not including tumor biopsy, ablation therapy, etc.) within 2 weeks before trial drug treatment;
3. Adverse events from previous anti-tumor treatments have not recovered to ≤ grade 1 according to CTCAE v5.0 (except for ≤ grade 2 toxicities judged by the investigator to have no safety risk, such as alopecia, long-term toxicity caused by radiotherapy, etc.);
4. Patients with known brain metastases. Those with stable brain metastases can be enrolled;
5. Third space effusion that is clinically uncontrollable and unsuitable for enrollment;
6. Participants with≥ grade 3 allergies to antibody drugs previously;
7. Taking systemic corticosteroids (>10 mg daily prednisone or equivalent dose) or other systemic immunosuppressive drugs (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate , thalidomide, and anti-tumor necrosis factor drugs), topical, ocular, intra-articular, intranasal, and inhaled corticosteroids are allowed;
8. Subjects with a known history of autoimmune diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, Guillain-Barre syndrome, multiplex syndrome sclerosis or glomerulonephritis, except autoimmune-related hypothyroidism treated with stable dose of hormone;
9. Known idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonia, idiopathic pneumonia, interstitial lung disease, severe radiation pneumonitis, or subjects with evidence of active pneumonia by chest CT scan screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 weeks
  Objective Response Rate

SECONDARY OUTCOMES:
DoR | 6 weeks
  Duration of overall response
DCR | 6 weeks
  Disease control rate
PFS | 6 weeks
  Progression-free survival
OS | 6 weeks
  Overall survival
Adverse events | 6 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China